CLINICAL TRIAL: NCT07080554
Title: "Analysis of Diagnostic Criteria for Primary Sarcopenia in Community-dwelling Older Adults vs. Institutionalized in Nursing Homes"
Brief Title: Observational and Analytical Study on the Diagnostic Criteria for Sarcopenia in Institutionalized Older Adults and Those Living in the Community
Status: Completed | Type: Observational
Sponsor: University of Extremadura (Other)
Responsible Party: Principal Investigator, Jesús Zapata Linares, Clinical professor, University of Extremadura
Other Study IDs: 01
Record Dates: First submitted 2025-06-28; First posted 2025-07-23 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-07

CONDITIONS: Sarcopenia in Elderly; Institutionalized Older Adults; Community-dwelling Elderly

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- This group includes institutionalized older adults aged 60 and over.
- This group includes community-dwelling older adults aged 60 and over.

SUMMARY:
Sarcopenia is one of the main problems in the elderly population. However, its diagnostic criteria have not yet been studied in two specific populations, namely institutionalized older adults in nursing homes vs community-dwelling older adults. So this will be the objective of the study. An observational study is being conducted to analyze how these diagnostic criteria relate to each other and to find possible associations.

ELIGIBILITY:
Inclusion Criteria:

* older adults who have been institutionalized for at least one year
* older adults who are institutionalized with clinical suspicion of sarcopenia according to the Sarc-F questionnaire and muscle strength criteria
* older adults residing in the community of Extrema

Exclusion Criteria:

* present cognitive impairment (score <24 Mini-Mental State Examination)
* primary, serious, or chronic diseases that could explain the decrease in muscle strength and the other diagnostic variables of the participants
* diseases or physical disorders that hinder the assessment of the participants; -use of drugs that may affect muscle strength and mass [35].

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study will include two groups: one group of institutionalized older adults in nursing homes with clinical sospicius of sarcopenia and another group of community-dwelling older adults apparently healthy.
Sampling Method: Non-Probability Sample
Enrollment: 415 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2024-02-01 (Actual)

PRIMARY OUTCOMES:
Hand grip strenght | Once at the baseline
  The researchers used the JAMAR dynamometer

SECONDARY OUTCOMES:
Muscular mass / appendicular skeletal mass (ASM) | Once at the baseline
  The researchers used bioimpedance analysis with Tanita MC780-S MA Multifrequency.
Physical performance | Once at the baseline
  The researchers used the scale: "Short Physical Performance Battery" (SPPB),
Physical performance 2 | Once at the baseline
  The researchers used the test: "Timed Up and Go" (TUG)

CONTACTS AND LOCATIONS:
Overall Officials: Luis Espejo-Antunez, Study Director — University of Extremadura
Locations (1):
- Universidad de Extremadura, Badajoz, Badajoz, Spain